CLINICAL TRIAL: NCT02272023
Title: Randomized Trial of Intensive Motivational Interviewing (IMI) to Improve Drinking Outcomes Among Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Institute, California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AA022857 (NIH)
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Alcohol Use Disorders
Keywords: alcohol; women; motivational interviewing
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 9 sessions of Intensive Motivational Interviewing (Experimental): Experimental condition will consist of 9 1-hour intensive motivational interviewing sessions.
  Interventions: Behavioral: Intensive Motivational Interviewing
- 1 Standard Motivational Interview plus 8 nutrition classes (Active Comparator): The standard MI intervention will consist of a commonly used, single session of MI (50 minutes) plus 8 hours of nutrition education to achieve time and attention equivalence of study conditions.
  Interventions: Behavioral: Single session of Motivational Interviewing

INTERVENTIONS:
Behavioral: Intensive Motivational Interviewing — Weekly individual therapy sessions over 9 weeks (Intensive MI condition) consisting of supportive and directive interventions. The control condition consists on a single session of MI and nutritional education.
  Arms: 9 sessions of Intensive Motivational Interviewing
Behavioral: Single session of Motivational Interviewing
  Arms: 1 Standard Motivational Interview plus 8 nutrition classes

SUMMARY:
A Phase II Randomized Clinical Trial (RCT) is proposed to compare a 9-session model of intensive motivational interviewing (IMI) to standard motivational interviewing techniques (SMI) among alcohol dependent women. Preliminary work studying 87 women randomly assigned to IMI or a standard single session of motivational interviewing showed significantly better drinking outcomes for women in the IMI condition at 4- and 6-month follow-up. Interestingly, mean trajectories for women assigned to IMI showed continuing declines in drinking problems during and after treatment. Differences between study conditions grew larger between 4-month (p<.05) and 6-month (p<.01) follow-up and the effect size at 6 months was medium to large (Cohen's d=0.63) The study will use mixed model quantitative and qualitative methods to respond to the PA's call for studies assessing mechanisms of change. Unlike many previous studies of SMI, we will employ limited exclusion criteria and will enroll participants who present with co-existing drug and psychiatric disorders.

Procedures for the proposed study draw from our current successful RCT assessing IMI for methamphetamine (MA) dependence. Successful aspects of the current study include achievement of recruitment goals, strong adherence to the treatment and research protocols, and excellent rates for follow-up interviews (>90%). The proposed study will take place at the same outpatient treatment program as the current study, New Leaf Treatment Center in Lafayette, California.

Participants will include 220 alcohol dependent women who will be randomly assigned to IMI or SMI. Those in SMI will also receive an attention component (nutrition education) to achieve time equivalence between the two study conditions. Participants in both groups will receive standard weekly group treatment offered at the program. In addition, referrals to Alcoholics Anonymous will be provided to all participants. The primary outcomes will be measures of drinking, heavy drinking (4+ drinks), and severity of alcohol problems assessed at baseline and 2, 6, and 12 months. Secondary outcomes will include Addiction Severity Index scales, psychiatric problems, and symptoms of trauma. The study will include standard quantitative testing of potential mediators, including, the therapeutic alliance, self-efficacy, motivation, satisfaction, and use of outside services. However, the application also proposes an innovative use of qualitative procedures to identify unrecognized factors influencing outcome.

DETAILED DESCRIPTION:
The proposed study responds to the Program Announcement PA-10-100, "Alcohol Use Disorders: Treatment, Services Research, and Recovery" (R01) issued by the National Institute on Alcohol Abuse and Alcoholism (NIAAA). Our application addresses the priorities of this announcement by proposing a phase II randomized clinical trial comparing intensive motivational interviewing (IMI) to standard motivational interviewing techniques (SMI) for alcohol dependent women. The study will use mixed model quantitative and qualitative methods to respond to the program announcement's call for studies assessing mechanisms of change. Unlike many previous studies of SMI we will employ limited exclusion criteria and will enroll participants who present with co-existing drug and psychiatric disorders.

SMI was initially developed as a brief intervention (typically 1-3 sessions) for the treatment of problem drinkers (Miller & Rollnick, 2002). The general strategy of SMI is to strategically combine supportive and directive interventions as a way to elicit ambivalence about substance use (i.e., pros and cons) and thereby increase motivation for change. Systematic reviews of the alcohol treatment literature have consistently shown SMI to be effective for treating alcohol use disorders (Hettema, Steele, & Miller, 2005; Dunn, Deroo, Rivera, 2001). Studies have shown SMI to be effective as a stand-alone treatment for alcohol problems (Project MATCH Research Group, 1997; Miller, 1993; Sellman, Sullivan, Dore, Adamson, & MacEwan, 2001) and as preparation for more intensive treatment (Burke, Arkowitz, & Menchola, 2003). Perhaps the best-known and largest study of an SMI based was an assessment of "motivational enhancement therapy" (MET) as a stand-alone, 4 session condition conducted by the Project MATCH Research Group (Sellman, Sullivan, Dore, Adamson, & MacEwan, 2001; Project MATCH Research Group, 1998). Participants were randomly assigned to 4 sessions of MET, 12 sessions of cognitive behavioral counseling (CBT), or 12 sessions of 12-step facilitation (TSF). Despite fewer sessions in MET, outcomes among the 3 conditions were comparable. A limitation of the study was that individuals with serious co-occurring drug or mental health problems were excluded as were those with housing instability.

Like Project MATCH, most studies of SMI for alcohol problems have excluded participants who have serious co-occurring drug and mental health problems. However, these are precisely the types of individuals that treatment practitioners are likely to encounter in publicly funded treatment programs. When SMI interventions have targeted illicit drug dependence the results have been mixed. While a number of reviews (Dunn, Deroo, Rivera, 2001) and meta-analyses (Burke, Arkowitz, & Menchola, 2003; Hettema, Steele, & Miller, 2005) have concluded standard low-dose SMI is effective as preparation for more intensive drug treatment, some studies contradict these findings (Downey, Rosengren, & Donovan, 2001; Miller, Yahne, Tonigan, 2003; Winhusen et al., 2008; Mullins, Suerez, Ondersman, Page, 2004; Schneider, Casey, Kohn, 2000). When effects have been found for drug and co-occurring disorders they have most commonly been for retention, not substance use (Carroll et al., 2006).

Procedures for the proposed study draw from our current successful RCT assessing IMI for MA dependence. Successful aspects of the current study include achievement of recruitment goals, strong adherence to the treatment and research protocols, and excellent rates for follow-up interviews (>90%). The proposed study will take place at the same outpatient treatment program as the current study, New Leaf Treatment Center in Lafayette, California. Two hundred and twenty alcohol dependent women will be randomly assigned to IMI or SMI with an attention component for time equivalence (nutrition education). Participants in both groups will receive standard group treatment offered at the program. The primary outcomes will be measures of drinking, heavy drinking (4+ drinks), and severity of alcohol problems assessed at baseline and 2, 6, and 12 months. Secondary outcomes will include Addiction Severity Index scales, psychiatric problems, and symptoms of trauma. The study will include standard quantitative testing of potential mediators, including, the therapeutic alliance, self-efficacy, motivation, satisfaction, and use of outside services. However, the application also proposes an innovative use of qualitative procedures to identify unrecognized factors influencing outcome.

Aim 1: To compare drinking and alcohol problems among women receiving IMI and SMI.

Hypothesis 1.1: During the active phase of treatment (weeks 1-9) women in IMI will have fewer positive breathalyzer screens, drinking days, and heavy drinking days (4+ drinks) than women in SMI.

Hypothesis 1.2: Women in IMI will demonstrate fewer drinking days and heavy drinking days (4+ drinks) and lower scores on the Addiction Severity Index (ASI) Alcohol Scale at 2, 6, and 12 months.

Aim 2: To assess potential mediators of drinking and alcohol problems. Hypothesis 2.1: Measures of retention, therapeutic alliance, social support, and motivation will mediate the relationship between study condition and drinking outcome.

Aim 3: To Use qualitative interviews to identify additional factors that influence outcome. Content areas will include perceptions of the therapist, IMI & SMI interventions, the CBT group, and external influences such as Alcoholics Anonymous (AA), intimate partners, friends, and family.

Exploratory Aims: 1) To compare IMI and SMI outcomes on ASI scales, psychiatric symptoms, AA involvement, and trauma symptoms.

ELIGIBILITY:
Inclusion Criteria:

1) Female 2)18 years or older 3) meets DSM-V criteria for current alcohol use disorder in the past 30 days, as assessed by the DSM-V Checklist, defined as 2 or more criterion 4) alcohol in the past 30 days and medically cleared by NLTC medical personnel 5) able to speak and read English, 6) capable of giving informed consent 7) likely to be in the area the next 12 months.

Exclusion Criteria:

1. has had alcohol in the past 3 days and may require medical treatment for alcohol or drug detoxification and is not followed by a physician or has not been medically cleared by NLTC medical personnel
2. or has unmet needs for treatment of serious medical or psychiatric conditions
3. any condition that would impair their ability to provide informed consent
4. current severe drug use disorder, defined as 6 or more DSM-V criteria in the past 30 days, 5.)Currently enrolled in alcohol or drug treatment

6) Does not meet DSM-V criteria for current alcohol use disorder as assessed by the DSM-V Checklist, 7) Refuses to sign HIPPA authorization form 8) Any medical or psychosocial condition that would preclude safe, useful, or consistent participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Change in the number of drinks and frequency of drinks in the past two months | Baseline, 2 months, 6 months, and 12 months
  Change in daily drinking patterns (quantity and frequency) over the past two months using the Timeline follow-back assessment
Change in the severity of alcohol use within past 30 days | Baseline, 2 months, 6 months, and 12 months
  Change in alcohol Addiction Severity Index (ASI) scores in the past 30 days

SECONDARY OUTCOMES:
Change in employment, psychiatric status, and legal status over the past 30 days | Baseline, 2 months, 6 months, and 12 months
  Change in employment, psychiatric status, and legal status over the past 30 days as assessed by the Addiction Severity Index (ASI)
Change in mental health | Baseline, 2 months, 6 months, and 12 months
  Change in emotions, moods, thoughts, and behaviors in the past two weeks as assessed by the Psychiatric Diagnostic Screening Questionnaire (PDSQ)
Change in trauma and stress levels | Baseline, 2 months, 6 months, and 12 months
  Change in drinking consequences scores as assessed by Alcohol and Drug Consequences Questionnaire (ADCQ)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Polcin, Ed.D., Principal Investigator — Alcohol Research Group / Public Health Institute
Locations (1):
- New Leaf Treatment Center, Lafayette, California, United States

REFERENCES:
- [Background] Burke BL, Arkowitz H, Menchola M. The efficacy of motivational interviewing: a meta-analysis of controlled clinical trials. J Consult Clin Psychol. 2003 Oct;71(5):843-61. doi: 10.1037/0022-006X.71.5.843. PMID 14516234
- [Background] Carroll KM, Ball SA, Nich C, Martino S, Frankforter TL, Farentinos C, Kunkel LE, Mikulich-Gilbertson SK, Morgenstern J, Obert JL, Polcin D, Snead N, Woody GE; National Institute on Drug Abuse Clinical Trials Network. Motivational interviewing to improve treatment engagement and outcome in individuals seeking treatment for substance abuse: a multisite effectiveness study. Drug Alcohol Depend. 2006 Feb 28;81(3):301-12. doi: 10.1016/j.drugalcdep.2005.08.002. Epub 2005 Sep 28. PMID 16169159
- [Background] Downey L, Rosengren DB, Donovan DM. Sources of motivation for abstinence: a replication analysis of the reasons for quitting questionnaire. Addict Behav. 2001 Jan-Feb;26(1):79-89. doi: 10.1016/s0306-4603(00)00090-3. PMID 11196294
- [Background] Dunn C, Deroo L, Rivara FP. The use of brief interventions adapted from motivational interviewing across behavioral domains: a systematic review. Addiction. 2001 Dec;96(12):1725-42. doi: 10.1046/j.1360-0443.2001.961217253.x. PMID 11784466
- [Background] Hettema J, Steele J, Miller WR. Motivational interviewing. Annu Rev Clin Psychol. 2005;1:91-111. doi: 10.1146/annurev.clinpsy.1.102803.143833. PMID 17716083
- [Background] Miller WR, Yahne CE, Tonigan JS. Motivational interviewing in drug abuse services: a randomized trial. J Consult Clin Psychol. 2003 Aug;71(4):754-63. doi: 10.1037/0022-006x.71.4.754. PMID 12924680
- [Background] Mullins SM, Suarez M, Ondersma SJ, Page MC. The impact of motivational interviewing on substance abuse treatment retention: a randomized control trial of women involved with child welfare. J Subst Abuse Treat. 2004 Jul;27(1):51-8. doi: 10.1016/j.jsat.2004.03.010. PMID 15223094
- [Background] Matching Alcoholism Treatments to Client Heterogeneity: Project MATCH posttreatment drinking outcomes. J Stud Alcohol. 1997 Jan;58(1):7-29. PMID 8979210
- [Background] Matching alcoholism treatments to client heterogeneity: Project MATCH three-year drinking outcomes. Alcohol Clin Exp Res. 1998 Sep;22(6):1300-11. doi: 10.1111/j.1530-0277.1998.tb03912.x. PMID 9756046
- [Background] Schneider RJ, Casey J, Kohn R. Motivational versus confrontational interviewing: a comparison of substance abuse assessment practices at employee assistance programs. J Behav Health Serv Res. 2000 Feb;27(1):60-74. doi: 10.1007/BF02287804. PMID 10695241
- [Background] Sellman JD, Sullivan PF, Dore GM, Adamson SJ, MacEwan I. A randomized controlled trial of motivational enhancement therapy (MET) for mild to moderate alcohol dependence. J Stud Alcohol. 2001 May;62(3):389-96. doi: 10.15288/jsa.2001.62.389. PMID 11414349
- [Background] Winhusen T, Kropp F, Babcock D, Hague D, Erickson SJ, Renz C, Rau L, Lewis D, Leimberger J, Somoza E. Motivational enhancement therapy to improve treatment utilization and outcome in pregnant substance users. J Subst Abuse Treat. 2008 Sep;35(2):161-73. doi: 10.1016/j.jsat.2007.09.006. Epub 2008 Feb 20. PMID 18083322
- [Background] Miller WR. What really drives change? Addiction. 1993 Nov;88(11):1479-80. doi: 10.1111/j.1360-0443.1993.tb03133.x. No abstract available. PMID 8286993
- See also: website — http://www.arg.org